CLINICAL TRIAL: NCT06248606
Title: Phase II Study of Adagrasib + Stereotactic Radiosurgery (SRS) for Patients With Metastatic KRAS G12C-mutated NSCLC With Untreated Brain Metastases
Brief Title: Adagrasib + SRS for Patients With Metastatic KRAS G12C-mutated NSCLC With Untreated Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ryan Gentzler, MD (Other)
Collaborators: Mirati Therapeutics Inc. (Industry); University of Virginia (Other)
Responsible Party: Sponsor-Investigator, Ryan Gentzler, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN LUN23-618
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer; NSCLC; KRAS G12C
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — adagrasib; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Adagrasib + SRS (Stereotactic Radiosurgery) (Experimental): All patients will receive oral adagrasib 600mg twice daily for every cycle and SRS which will be administered as standard of care. SRS will occur between 4 weeks prior to and up to 3 weeks after initiation of adagrasib. Patients may have received SRS prior to study enrollment. Cycle 1 Day 1 will begin on the first day of adagrasib dosing. Adagrasib should be held the day before and the day of SRS. There is no maximum duration of treatment.
  Interventions: Drug: Adagrasib; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Drug: Adagrasib — Adagrasib 600mg orally
  Other Names: Krazati
Radiation: Stereotactic Radiosurgery — Delivered as per standard of care
  Other Names: SRS

SUMMARY:
This is a single arm phase 2 trial is to evaluate the efficacy of SRS plus adagrasib for the treatment of brain metastases for patients with KRAS G12C-mutated non-small cell lung cancer (NSCLC). A total of 30 patients will be enrolled on this study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. ECOG Performance Status of 0-1 within 28 days prior to registration.
4. Confirmation of stage IV non-small cell lung cancer (NSCLC) per AJCC, 8th edition, or metastatic recurrence after treatment for earlier stage disease.
5. Known to have a KRAS G12C mutation. KRAS G12C mutation can be determined based on local tissue and/or ctDNA testing.
6. Presence of brain metastases that meet the following criteria:

   * Patients must have at least 1 untreated enhancing intracranial lesion, per local radiology interpretation, measuring at least 2mm. NOTE: intracranial lesions do not need to be measurable by RECIST 1.1 criteria to be eligible.
   * Must have no single metastasis measuring larger than 3 cm.
   * Patients with surgically resected brain metastases are eligible provided there are additional brain metastases amenable to SRS
   * Patients with progression of previously radiated or surgically resected CNS metastases are eligible if solid component of lesion has enlarged and there is no concern for radionecrosis based on investigator discretion.
   * Patients who received SRS within 4 weeks prior to registration are eligible provided baseline brain MRI prior to SRS treatment is within 4 weeks of study registration and SRS treatment meets requirements in #7 below.
   * Symptomatic brain metastases are permitted if the following criteria are met:

     * No evidence of cerebral herniation or symptomatic leptomeningeal disease
     * No seizures within past 14 days; antiepileptic medications are permitted
     * Patients on steroids must have stable or improving neurologic symptoms that have not worsened during a steroid taper. Must be receiving the equivalent of dexamethasone 8 mg total daily dose or less at the time of registration.
7. CNS lesions have already been treated with SRS (within 3 weeks prior to Cycle 1 Day 1) or are amenable to SRS as determined by radiation oncologist and/or neurosurgeon. SRS treatment must use GammaKnife or linear accelerator-based treatments with nominal x-ray energy of 6MV or greater.
8. No contraindications to SRS. Patients on anticoagulation must be able to hold anticoagulation for SRS treatment based on investigator discretion.
9. Patients may be treatment-naïve OR have received up to 2 prior lines of systemic therapy. Treatment with systemic therapy for Stage I-III disease > 12 months prior to development of metastases do not count as a line of therapy. Treatment with platinum-doublet chemotherapy and checkpoint inhibitor immunotherapy (PD-1, PD-L1, CTLA-4, etc.) either in combination or sequentially counts as one line of therapy.
10. Demonstrate adequate organ function as defined below. All screening labs to be obtained within 28 days prior to registration.

    * Hemoglobin (Hgb): ≥ 8.0 g/dL in the absence of transfusions within 7 days prior to testing.
    * Calculated creatinine clearance: ≥ 60 mL/min
    * Bilirubin: ≤ 1.5 mg/dL
    * Aspartate aminotransferase (AST): ≤ 3.0 × ULN
    * Alanine aminotransferase (ALT): ≤ 3.0 × ULN
11. Females of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to treatment initiation.
12. Females of childbearing potential who are sexually active with a male able to father a child must be willing to abstain from heterosexual activity or to use an effective method(s) of contraception. Males able to father a child who are sexually active with female of childbearing potential must be willing to abstain from heterosexual activity or to use an effective method(s) of contraception.
13. HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial. Testing is not required at screening unless mandated by local policy.
14. Patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, the HCV viral load must be undetectable to be eligible for this trial. Testing is not required at screening unless mandated by local policy.
15. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

1. Prior treatment with KRAS G12C tyrosine kinase inhibitor.
2. Active infection requiring systemic therapy with the exception of #13 and #14 above.
3. Uncontrolled, significant intercurrent or recent illness.
4. Prolonged QTc interval > 480 milliseconds or history of congenital Long QT Syndrome
5. Currently receiving radiation treatment at the time of enrollment to any extra-cranial lesion for prophylaxis or pain control. Patients may enroll after completion of palliative RT.
6. Ongoing need for treatment with concomitant medication known as a strong inhibitor or inducer of CYP3A enzyme and that cannot be switched to an alternative treatment prior to study enrollment. NOTE: Discontinuation of CYP3A4 inducers should occur a minimum of 7 days or 5 times their half-life, whichever is longer, prior to C1D1 study treatment.
7. Treatment with any investigational drug within 28 days prior to registration.
8. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
9. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen, per treating physician discretion, are not eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Intracranial disease control rate (DCR) | 3 months
  Intracranial disease control rate (DCR) [complete response (CR) + partial response (PR) + stable disease (SD)] per RECIST 1.1 for intracranial lesions at 3 months

SECONDARY OUTCOMES:
Adverse events | 52 months
  Safety and tolerability will be assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).
Intracranial overall response rate (ORR) | 52 months
  Intracranial overall response rate (icORR) will be measured by RECIST 1.1 criteria including only intracranial lesions. icORR is defined as the proportion of patients who have a partial or complete response (PR or CR) to therapy for intracranial lesions.
Overall response rate (ORR) | 52 months
  ORR will be measured by RECIST 1.1. ORR is defined as the proportion of patients who have a partial or complete response to therapy for all disease (systemic and intracranial lesions).
Progression free survival (PFS) | 52 months
  PFS is defined as time from the day of study treatment initiation until evidence of disease progression at any location per RECIST v1.1, or death from any cause.
Overall survival (OS) | 52 months
  OS will be calculated starting from the day of study treatment initiation until death from any cause.
Intracranial progression free survival (PFS) | 52 months
  Intracranial PFS is defined as time from the day of study treatment initiation until evidence of disease progression in the brain per RECIST 1.1 criteria including only intracranial lesions or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Gentzler, MD, MS, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia